CLINICAL TRIAL: NCT05544864
Title: Intracoronary Stenting and Restenosis - Randomized Trial of Drug-eluting Stent Implantation or Drug-coated Balloon Angioplasty According to Neointima Morphology in Drug-eluting Stent Restenosis 5
Acronym: ISAR-DESIRE5
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: EvidentIQ Germany GmbH (Unknown); Abbott (Industry); Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE no. BA00219
Record Dates: First submitted 2022-09-09; First posted 2022-09-19 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Coronary Artery Disease; Restenoses, Coronary
MeSH Terms: conditions — Coronary Artery Disease; Coronary Restenosis | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- homogenous (Other): Stratification - homogenous pattern
  Interventions: Device: Drug eluting stent (DES); Device: Drug coated ballloon (DCB)
- heterogenous (Other): Stratification - homogenous pattern
  Interventions: Device: Drug eluting stent (DES); Device: Drug coated ballloon (DCB)

INTERVENTIONS:
Device: Drug eluting stent (DES) — DES-implantation with an everolimus-eluting stent (Xience, Abbott Vascular)
Device: Drug coated ballloon (DCB) — DCB angioplasty with any commercially available drug-coated balloon

SUMMARY:
The hypothesis of the study is, that there is a significant interaction in treatment effect between the OCT pattern of neointima (heterogeneous or homogeneous) and the type of percutaneous coronary intervention (drug-eluting stent or drug-coated balloon) in patients with in-stent restenosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ischemic symptoms and/or evidence of myocardial ischemia
2. Presence of ≥ 50% restenosis after prior implantation of drug-eluting stents in native coronary vessels.
3. Availability of an OCT-pullback of the target lesion
4. Written informed consent by the patient for participation in the study.
5. Age ≥ 18 years

Exclusion Criteria:

1. Cardiogenic shock
2. Acute ST-elevation myocardial infarction within 48 hours from symptom onset.
3. Target lesion located in left main trunk or bypass graft.
4. Additional coronary intervention planned within 30 days of the procedure.
5. Non-successful treatment of other lesion(s) during the same procedure
6. Severe renal insufficiency (glomerular filtration rate ≤ 30 ml/min)
7. Contraindications to any components of the investigational devices or dual antiplatelet therapy
8. Pregnancy (present, suspected or planned) or positive pregnancy test.
9. Previous enrollment in this trial or participation in any other study at the time of enrollment.
10. Malignancies or other comorbid conditions with life expectancy less than 12 months or that may result in protocol non-compliance.
11. Patient's inability to fully comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of major adverse cardiac event (MACE) | 24 months of clinical follow-up after randomization
  Composite endpoint of major adverse cardiac event (MACE)
  * all-cause death
  * myocardial infarction
  * target lesion revascularization (TLR)

SECONDARY OUTCOMES:
Target lesion failure (TLF): a composite of cardiac death, target-vessel myocardial infarction and TLR | 24 months of clinical follow-up after randomization
Individual endpoints of the composite endpoints | 24 months of clinical follow-up after randomization
  * all-cause death
  * myocardial infarction
  * target lesion revascularization (TLR)
Stent thrombosis according to the ARC criteria | 24 months of clinical follow-up after randomization
Safety endpoint: a composite endpoint of all-cause death and myocardial infarction | 24 months of clinical follow-up after randomization

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (4):
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Elisabeth-Krankenhaus Essen GmbH, Essen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Deutsches Herzzentrum München, Munich
- Hospital Universitario de La Princesa Madrid, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Simonetti F, Voll F, Alfonso F, Grasser C, Janisch M, Joner M, Kessler T, Kuna C, Leistner DM, Lenz T, Presch A, Rheude T, Sager H, Schunkert H, Starnecker F, Wiebe J, Kastrati A, Cassese S, Xhepa E. Intracoronary Stenting and Restenosis - Randomized Trial of Drug-Eluting Stent Implantation or Drug-Coated Balloon Angioplasty According to Neointima Morphology in Drug-Eluting Stent REstenosis 5: Rationale and Design of the ISAR-DESIRE 5 Trial. J Cardiovasc Transl Res. 2025 Oct;18(5):1176-1184. doi: 10.1007/s12265-025-10650-x. Epub 2025 Jun 30. PMID 40588613